CLINICAL TRIAL: NCT04581161
Title: A Novel Proportional Open Ventilation (POV) Device and Its Efficacy in Managing Acute Respiratory Failure in COVID-19 Patients
Brief Title: Proportional Open Ventilation (POV) Device and Its Efficacy in Managing Acute Respiratory Failure in COVID-19 Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hill-Rom (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR-RR-2020-004
Record Dates: First submitted 2020-08-19; First posted 2020-10-09 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Acute Respiratory Failure; Covid19
Keywords: ARDS; PEEP; Respiratory Rate
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Subjects in the active treatment group will receive ventilatory support with Life2000® Ventilator following the labeled instructions for the device.
  POV support (Life2000) will be administered in six (6) to ten (ten) enrolled subjects based on clinical protocol flowchart (Appendix C). Specifically, if it is determined that a COVID-19 subject who would currently be considered for HFNC under current standard of treatment, will be eligible for POV treatment.
  The prescribed therapy regimen, including duration of therapy will be documented and COVID-19 patients who fail therapy and require IMV will be recorded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Life2000® Ventilator (Experimental): Subjects in the active treatment group will receive ventilatory support with Life2000® Ventilator following the labeled instructions for the device.
  Interventions: Device: Life2000® Ventilator
- Control Group (No Intervention): Subjects in the control group will be identified from the population of patients previously admitted to the study site with COVID-19 infection who required non-invasive oxygen therapy with HFNC but were not treated with NIV therapy. Subject data will be collected retrospectively from the medical record.

INTERVENTIONS:
Device: Life2000® Ventilator — POV support (Life2000) will be administered in six (6) to ten (ten) enrolled subjects based on clinical protocol flowchart (Appendix C). Specifically, if it is determined that a COVID-19 subject who would currently be considered for HFNC under current standard of treatment, will be eligible for POV treatment.
  The prescribed therapy regimen, including duration of therapy will be documented and COVID-19 patients who fail therapy and require IMV will be recorded.
  Arms: Life2000® Ventilator

SUMMARY:
To evaluate the use of Life2000® Ventilator, a novel proportional open ventilation system in critical care use of acute onset of respiratory failure (ARF) and mild to moderate forms of acute respiratory distress syndrome (ARDS) in COVID-19 patients and its ability to provide effective ventilatory benefits and or delay patients from progressing to more aggressive forms of invasive mechanical ventilation (IMV).

ELIGIBILITY:
Inclusion Criteria:

Patients who meet all of the following inclusion criteria and no exclusion criteria will be included in the study:

* A diagnosed or suspected COVID-19 patient requiring non-invasive ventilatory support and admitted to hospital
* PaO2/FiO2 ≤ 300 (corrected for altitude)
* RR ≤ 30/min during early use of oxygen
* Adults of 18 years and older
* Provision of written informed consent to participate in study by subject or legal representative.

Exclusion Criteria:

Patients who meet one or more of the following exclusion criteria will not be eligible for the study:

* Patients under the age of 18
* Patients who are not diagnosed or suspected of having an acute COVID-19 illness
* Patients who do not require non-invasive ventilatory interventions, PaO2/FiO2 > 300 (corrected for altitude) and tolerating supplemental oxygen with SpO2 saturations ≥ 92%.
* Patients who require immediate IMV upon admission or have a RR > 30/min on early oxygen intervention.
* Thoracoabdominal desynchrony and paradoxical breathing at admission
* Patients in immediate need of or on vasopressors upon ICU admission
* Patients or legal representatives who are unwilling or unable to provide written consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-08-28 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Life2000® Compared to HFNC (AIRVO) | Time frame measured will include date that patient is admitted to hospital until date patient is discharged from hospital or death occurs with an anticipated 30 day time period, but shall not exceed 90 day time period.
  Compared to HFNC (AIRVO), does the Life2000® Ventilator provide clinically relevant ventilatory support to COVID-19 patients with mild to moderate ARF or ARDS to prevent IMV.

SECONDARY OUTCOMES:
PEEP level | Time frame measured will include date that patient is admitted to hospital until date patient is discharged from hospital or death occurs with an anticipated 30 day time period, but shall not exceed 90 day time period.
  What level of PEEP is required to ensure adequate ventilation in COVID-19 patients with mild to moderate ARF/ARDS.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Shelver, MD, Principal Investigator — Park Nicolette
Locations (1):
- Park Nicolette, Bloomington, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No